CLINICAL TRIAL: NCT01461070
Title: BRANCH:Fecal Microbiota Among Participants in a Pre-paid Health Plan
Brief Title: Intestine Bacteria and Breast Cancer Risk
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911235; 11-C-N235
Record Dates: First submitted 2011-10-06; First posted 2011-10-27 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Breast Neoplasms
Keywords: Breast Cancer; Post Menopausal Estrogens; Fecal Microbes
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Feces and urine.

GROUPS / COHORTS (2):
- Breast Cancer Cases: Breast Cancer Cases
- Controls: Controls

SUMMARY:
Background:

- Some bacteria found in the large and small intestines help keep people healthy and aid digestion. They may also affect a person s risk of developing cancer. Researchers want to study the relationship between intestinal bacteria and breast cancer risk factors. They can do this by looking at stool and urine samples from postmenopausal women.

Objectives:

- To study intestinal bacteria and its relationship to urine-based markers of breast cancer risk in women.

Eligibility:

- Women between 55 and 69 years of age with a recent mammogram that showed no signs of cancer.

Design:

* Participants will be screened with a medical history and basic health questionnaire.
* At home, participants will complete questionnaires about cancer risk factors and food consumption.
* Participants will also collect urine and stool samples. They will send the samples to the designated labs for study.
* No treatment will be provided as part of this protocol.

DETAILED DESCRIPTION:
Background/Significance: Commensal microbes (the microbiota), particularly in the gut, are required for human health and are postulated to affect cancer risk through several mechanisms. This proposed study builds upon a pilot within the NCI Division of Cancer Epidemiology and Genetics (DCEG) that identified highly acceptable methods for collecting fecal specimens and significant correlation between fecal microbial beta-glucuronidase activity and a marker of breast cancer risk, urine levels of estrogens. The proposed study will determine the correlation between levels of fecal enzyme activities and systemic estrogens in a random sample of postmenopausal women at Kaiser Permanente Colorado (KPCO). Demonstration of an association between the fecal microbiota and systemic estrogens would help to motivate future studies of how microbes affect cancer risk.

Objectives: The main objective is to characterize the fecal microbiota and its association with levels of systemic estrogens among randomly sampled postmenopausal female members of a health maintenance organization (HMO). A secondary objective will determine the proportions of women who consent and then provide questionnaire data, a fecal specimen to characterize the microbiota, and a urine specimen to quantify systemic estrogens; and differences between participants (N=60) and non-participants. A third objective will determine whether consecutive, newly diagnosed postmenopausal breast cancer cases have similar participation rates, fecal microbiota characteristics and urine estrogen levels compared to the randomly sampled women.

Methods: We will randomly sample from the KPCO population of approximately 50,000 women ages 55-69 who have recently had a negative screening mammogram. An invitation packet (letter, information pamphlet, consent form, eligibility questionnaire, and opt-out postcard) will be sent in batches of 100, up to a maximum of 500 women. The consenting women will receive a second packet with a cancer risk-factor questionnaire, a link to the on-line Block brief food frequency questionnaire, and a specimen collection kit (with illustrated instructions) for collecting a fecal and urine specimen. Participants (minimum 60, maximum 80) will ship the specimens to the DCEG repository. As amended, consecutive newly diagnosed breast cancer cases (target N=60) will be enrolled in the oncology clinic prior to definitive surgery, with the same eligibility criteria as for the random sample. For contemporaneous controls, participants in the randomly sampled, mammogram-negative population will be recruited back (target N=60). Urine estrogens will be quantified by DCEG at NCI Frederick. Fecal microbial classification and enzymatic expression and activity will be performed at the University of Maryland Medical School (UMMS).

Analyses: Data will be analyzed and summarized for publication with representatives from KPCO, DCEG and UMMS. Simple proportions will be used to estimate participation rates. Extant electronic records at KPCO will be used to compare participants to non-participants, overall and by pre-specified subgroups (5-year age groups, race/ethnicity, length of KPCO enrollment), with descriptive statistics and logistic regression. For the primary objective, fecal microbial 16S rRNA pyrosequences will be classified by phylogenetic and principal components analyses, while estrogen levels and Beta-glucuronidase RNA expression and enzymatic activity levels will be categorized using log standard deviations. The study will have 80% power to detect a 17% increase in estrogen level per 2.4-fold increase in glucuronidase activity and 80% power to detect a 3-fold case-control difference in above-median microbiome alpha diversity.

ELIGIBILITY:
* INCLUSION CRITERIA:

Female members of Kaiser Permanente Colorado (KPCO) with a recent normal mammogram who gets into a random sample of the very large population.

EXCLUSION CRITERIA:

History of cancer, except non-melanoma skin cancer

History of inflammatory bowel disease or diverticulitis

History of gastric banding or by-pass surgery

History of other gastric or intestinal surgery within the previous 6 months

Hormone prescription within the previous 12 months

Antibiotic prescription within the previous 6 months.

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Examining fecal microbiota in women with breast cancer
Sampling Method: Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2011-08-10 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
Breast cancer association | cross-sectional
  breast cancer association

SECONDARY OUTCOMES:
Fecal microbiome-systemic estrogen association | cross-sectional

CONTACTS AND LOCATIONS:
Overall Officials: Rashmi Sinha, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Kaiser Permanente Colorado, Denver, Colorado, United States

REFERENCES:
- [Background] Fuhrman BJ, Feigelson HS, Flores R, Gail MH, Xu X, Ravel J, Goedert JJ. Associations of the fecal microbiome with urinary estrogens and estrogen metabolites in postmenopausal women. J Clin Endocrinol Metab. 2014 Dec;99(12):4632-40. doi: 10.1210/jc.2014-2222. PMID 25211668
- [Background] Feigelson HS, Bischoff K, Ardini MA, Ravel J, Gail MH, Flores R, Goedert JJ. Feasibility of self-collection of fecal specimens by randomly sampled women for health-related studies of the gut microbiome. BMC Res Notes. 2014 Apr 1;7:204. doi: 10.1186/1756-0500-7-204. PMID 24690120
- [Background] Goedert JJ, Jones G, Hua X, Xu X, Yu G, Flores R, Falk RT, Gail MH, Shi J, Ravel J, Feigelson HS. Investigation of the association between the fecal microbiota and breast cancer in postmenopausal women: a population-based case-control pilot study. J Natl Cancer Inst. 2015 Jun 1;107(8):djv147. doi: 10.1093/jnci/djv147. Print 2015 Aug. PMID 26032724